CLINICAL TRIAL: NCT07173504
Title: The Effect of Continuous Versus Intermittent Enteral Nutrition on Metabolic Outcomes in Critically Ill Patients
Acronym: CONVEnIENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gelderse Vallei Hospital (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Wageningen University and Research (Other)
Responsible Party: Principal Investigator, ARH van Zanten, MD PhD, Internist-intensivist, Medical Head of ICU and Research, Gelderse Vallei Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL88158.091.24
Record Dates: First submitted 2025-08-05; First posted 2025-09-15 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Critical Illness
Keywords: critical illness; tube feeding; glycemic control; chrononutrition
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous enteral nutrition (No Intervention): Participants will receive the standard of care, continuous enteral nutrition for 24 hours a day.
- Intermittent enteral nutrition (Experimental): Participants will receive intermittent enteral nutrition in four separate portions between 8:00 a.m. and 8:00 p.m. Each portion will be administered over a one-hour period.
  Interventions: Other: Intermittent enteral nutrition

INTERVENTIONS:
Other: Intermittent enteral nutrition — Participants will receive intermittent enteral nutrition in four separate portions between 8:00 a.m. and 8:00 p.m. Each portion will be administered over a one-hour period.
  Other Names: Intermittent tube feeding
  Arms: Intermittent enteral nutrition

SUMMARY:
The goal of this clinical trial is to investigate the effect of continuous versus intermittent enteral nutrition on metabolic outcomes in critically ill adult patients.

The aim of this study is to:

• To assess the effect of a daytime intermittent tube feeding pattern compared to standard continuous tube feeding on glycaemic control, gastrointestinal function, gastrointestinal hormones, markers of sleep quality and circadian rhythm, and lean body mass and body composition.

Participants will receive either continuous enteral nutrition for 24 hours a day or intermittent enteral nutrition during the day, consisting of 4 portions each administered over 1 hour between 8 am and 8 pm. The maximum duration of the intervention is 5 days or until participants do not receive exclusive gastric enteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Receiving or eligible to receive exclusively gastric tube feeding;
3. Expected ICU stay ≥48 hours;
4. Receiving or anticipated to receive invasive mechanical ventilation within 48 hours after ICU admission.

Exclusion Criteria:

1. The treating clinician considers participation in the study clinically contraindicated (e.g., change in feeding regimen, no possibility for placement of CGM on arms, not able to receive exclusive gastric tube feeding);
2. Death is deemed to be imminent or inevitable during admission, and the attending doctor, patient, or substitute decision-maker is not committed to active treatment;
3. Pregnancy;
4. Expected fasting for ≥12 hours during the study period, for example, due to medical procedures;
5. Readmission in last 14 days;
6. Patients with burn injuries;
7. Participating in another nutritional intervention study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Glycaemic variability | From enrollment to the end of the intervention at a maximum of 5 days.
  The primary outcome is the mean glycaemic variability per 24 hours during the intervention, measured with Continuous Glucose Monitoring (CGM), expressed as the Coefficient of Variation (COV). The COV is calculated by dividing the standard deviation by the mean blood glucose level and multiplying by 100. It gives a relative measure of variability, which is helpful in comparing variability between individuals or groups with different mean glucose levels.

SECONDARY OUTCOMES:
Glycaemic control | From enrollment to the end of the intervention at a maximum of 5 days
  Assessed by mean and standard deviation of interstitial glucose concentrations and Mean Amplitude of Glycaemic Excursions (MAGE) (mmol/L)
Insulin administred during intervention period | From enrollment to the end of the intervention at a maximum of 5 days
  Insulin administred during intervention period (IU/day)
Dysglycemic events during intervention period | From enrollment to the end of the intervention at a maximum of 5 days
  Number of hypoglycaemic events, defined as blood glucose level <4.0 mmol/L and number of hyperglycaemic events, defined as blood glucose level >10.0 mmol/L
Gastrointestinal tolerance during the intervention period | From enrollment to the end of the intervention at a maximum of 5 days.
  Gastric residual volumes (mL), minimum, maximum and total volume per 24 hours.
Gastrointestinal tolerance during the intervention period | From enrollment to the end of the intervention at a maximum of 5 days
  Incidence of vomiting, diarrhoea, constipation and regurgitation during the intervetion periode
Circadian rhythm | Measured at day 1 and the end of the study period. End of the study period is day 5 of the study or earlier in case of: extubation, patient is no longer exclusively fed by gastric enteral nutrition or patient is discharged from ICU.
  Assessed by 24-hour curves of melatonin ( pg/mL) in saliva.
Circadian rhythm | Measured at day 1 and the end of the study period. End of the study period is day 5 of the study or earlier in case of: extubation, patient is no longer exclusively fed by gastric enteral nutrition or patient is discharged from ICU.
  Assessed by 24-hour curves of cortisol( nmol/L) in saliva.
Circadian rhythm | Measured at day 1 and the end of the study period. End of the study period is day 5 of the study or earlier in case of: extubation, patient is no longer exclusively fed by gastric enteral nutrition or patient is discharged from ICU.
  Assessed by 24-hour curves of mRNA expression of essential clock genes (BMAL, CLOCK, Cry1 and Per2).
Body composition | Measured at day 1 and the end of the study period. End of the study period is day 5 of the study or earlier in case of: extubation, patient is no longer exclusively fed by gastric enteral nutrition or patient is discharged from ICU.
  Fat-free mass, fat mass and skeletal muscle mass (kg and %) by bio-electrical impendence analysis. This outcome is only measured in centres with the necessary equipment.
Muscle size | Measured at day 1 and the end of the study period. End of the study period is day 5 of the study or earlier in case of: extubation, patient is no longer exclusively fed by gastric enteral nutrition or patient is discharged from ICU.
  Cross-sectional area and muscle layer thickness of quadriceps muscle by ultrasonography. This outcome is only measured in centres with the necessary equipment.
Nutritional intake during intervention period | From enrollment to the end of the intervention at a maximum of 5 days.
  Total nutritional prescription and delivery per calendar day (energy in kJ/day, protein in g/day, fat in g/day and carbohydrate in g/day and % of total intake)
Non-nutritonal calories administred during intervention period | From enrollment to the end of the intervention at a maximum of 5 days
  Non-nutritional calories delivered by propofol, glucose infusion, and citrate, delivery in kJ per calendar day
Health-related quality of life | 60 days after ICU admission
  Health-related quality of life measured with the 36-Item Short Form Health Survey (SF-36), 60 days after ICU admission
Sleep quality | 60 days after ICU admission
  Sleep quality measured with the Pittsburgh Sleep Quality Index (PSQI)
Glucoregulatory gastrointestinal hormones | From 12:00 until 14:00 on the second study day.
  GLP-1, C-peptide, insulin, and glucagon concentrations (mmol/L). This outcome is only measured in the coordinating centre.

OTHER OUTCOMES:
ICU length of stay | During index ICU stay, up to 60 days.
  ICU length of stay
Days on mechanical ventilation | During index ICU stay, up to 60 days.
  Days on mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Gelderse Vallei Hospital, Ede, Gelderland
  - Martini Ziekenhuis, Groningen, Provincie Groningen

IPD SHARING:
Plan to Share IPD: Undecided